CLINICAL TRIAL: NCT05640102
Title: A Phase 4, Observational Study Evaluating the Efficacy and Safety of the Bruton Tyrosine Kinase (BTK) Inhibitor Zanubrutinib in Patients With Waldenström Macroglobulinemia
Brief Title: Observational Study Evaluating the Efficacy and Safety of Zanubrutinib in Participants With Waldenström Macroglobulinemia
Status: Recruiting | Type: Observational
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Other Study IDs: BGB-3111-402
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-06

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: MYD88 L265P mutation: Arm A: Treatment-naïve (TN); Arm B: Relapsed/refractory (R/R)
  Interventions: Drug: Zanubrutinib
- Cohort 2: Non-L265P MYD88 mutation(s) and MYD88 wildtype: Arm C: TN and R/R
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Dosing and treatment duration are at the discretion of the prescribing physician and in accordance with local labeling
  Other Names: BGB-3111; Brukinsa

SUMMARY:
This is a hybrid (retrospective and prospective) non-interventional registry study to further describe the clinical profile of zanubrutinib in Waldenström macroglobulinemia (WM) participants with and without specific mutations and from racial and ethnic minority groups. Data collected from this registry study will be used to better understand the clinical benefit and safety of zanubrutinib for the treatment of participants in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and definitive histologic diagnosis of WM
* Measurable disease, as defined by a serum immunoglobulin M (IgM) level > 0.5 g/dL at the time of zanubrutinib initiation
* Started treatment with zanubrutinib, has been treated with zanubrutinib, or is planned to be prescribed zanubrutinib for the treatment of WM
* Bone marrow specimens with central MYD88 test results of:

  1. Cohort 1: MYD88 L265P mutation; enrollment of TN participants will be stopped in each racial and ethnic participant group when the required numbers of participants in the group are met
  2. Cohort 2: non-L265P MYD88 mutation(s) and MYD88WT

Exclusion Criteria:

* Evidence of disease transformation before the first dose of zanubrutinib
* Evidence of other non-Hodgkin Lymphoma (NHL) subtypes
* Prior or concurrent active malignancy ≤ 2 years before the first dose of zanubrutinib, except for malignancies that, in the investigator's opinion, will not obscure the interpretation of safety or efficacy results
* Concurrent participation in another therapeutic clinical study while receiving zanubrutinib, although the participant may be eligible depending on the status of the interventional study after discussion with the Medical Monitor or designee on an individual basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with WM who are either already receiving or are planned to start treatment with zanubrutinib
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Major Response Rate (MRR) | Up to approximately 4 years
  MRR is defined as the proportion of participants achieving either complete response (CR), very good partial response (VGPR), or partial response (PR) as determined by the investigator using an adaptation of the response criteria updated at the Sixth International Workshop on WM (IWWM)

SECONDARY OUTCOMES:
VGPR+ Rate | Up to approximately 5 years
  VGPR+ rate is defined as the proportion of participants achieving either CR or VGPR
Overall Response Rate (ORR) | Up to approximately 5 years
  ORR is defined as the proportion of participants achieving either CR, VGPR, PR, or minor response (MR)
Duration of Response (DOR) | Up to approximately 5 years
  DOR is defined as the time from the first determination of response (CR, VGPR, or PR) until first documentation of or death, whichever comes first
Number of Participants with Treatment-emergent Adverse Events | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (8):
- United States (7):
  - Clearview Cancer Institute, Huntsville, Alabama
  - South Alabama Medical Science Foundation Mitchell Cancer Institute, Mobile, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Los Angeles Cancer Network (Lacn), Glendale, California
  - Eisenhower Medical Center, Lucy Curci Cancer Center, Rancho Mirage, California
  - Hattiesburg Hematology and Oncology Clinic, Hattiesburg, Mississippi
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
- Pan American Oncology Trials, Llc, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/